CLINICAL TRIAL: NCT05504837
Title: KB407-02 A Phase 1 Study of Inhaled KB407, a Replication-Defective, Non-Integrating Vector Expressing Human Cystic Fibrosis Transmembrane Conductance Regulator, for the Treatment of Cystic Fibrosis
Brief Title: A Study Assessing KB407 for the Treatment of Cystic Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB407-02
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (open label) (Experimental): A single administration of KB407
  Interventions: Biological: KB407 (Nebulization)
- Cohort 2 (open label) (Experimental): Two administrations of KB407
  Interventions: Biological: KB407 (Nebulization)
- Cohort 3 (open label) (Experimental): Four administrations of KB407
  Interventions: Biological: KB407 (Nebulization)

INTERVENTIONS:
Biological: KB407 (Nebulization) — Nebulized solution of KB407, a replication-defective HSV-1 expressing full length human CFTR

SUMMARY:
This study will evaluate safety and tolerability of ascending doses of nebulized KB407 in adults with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have read, understood, and signed an Institutional Review Board/Ethics Committee (IRB/IEC) approved Informed Consent Form and must be able to and willing to follow study procedures and instructions
2. Subjects aged 18 years or older at the time of Informed Consent
3. A confirmed diagnosis of CF as defined by clinical signs and symptoms of CF and at least one of the following:

   * A historical sweat chloride value >60 mmol/L
   * Two copies of a disease causing mutation in the CFTR gene
4. Clinically stable in the opinion of the Investigator
5. Percent predicted FEV1 ≥40% and ≤100% of the predicted normal for age, gender, and height at Screening
6. Resting oxygen saturation ≥92% on room air at Screening

Exclusion Criteria:

1. Initiation of any new chronic therapy (eg, CFTR modulator, hypertonic saline, inhaled antibiotic) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days prior to the first dose
2. Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness 14 days prior to the first dose that, in the opinion of the Investigator, may confound study results
3. Treatment for Burkholderia cenocepacia, Burkholderia dolosa, or Nontuberculosis Mycobacteria infection within 3 months prior to the first dose
4. Participation in another clinical study or treatment with an investigational agent 30 days or 5 half-lives, whichever is longer, prior to the first dose
5. History of or listed for solid organ transplantation
6. Any condition (including a history or current evidence of substance abuse or dependence, uncontrolled asthma, or is considered to be immunocompromised) that, in the opinion of the Investigator, would impact a subject's ability to complete all study-related procedures and/or poses an additional risk to the assessment of safety of KB407
7. An active oral herpes infection 30 days prior to the first dose
8. Has received a vaccine within 72 hours prior to the first dose or has a planned vaccination during the treatment period
9. Women who are pregnant or nursing
10. Subject who is unwilling to comply with contraception requirements per protocol
11. Clinically significant abnormalities of hematology or chemistry testing at Screening that the Investigator believes may interfere with the assessment of safety and/or efficacy of the study treatment
12. Subject has a known hypersensitivity to inhaled glycerol
13. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the Investigator
14. Bronchoscopy participants only: Unable to tolerate bronchoscopy procedure and airway sampling, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of KB407 based upon assessment of adverse events (frequency, severity, relatedness), and changes from baseline in physical examinations, vital signs, ECG, and clinical laboratory test results | 2 months
  Number of adult subjects with treatment related adverse events as assessed by NCI-CTCAE v5

SECONDARY OUTCOMES:
To evaluate the effects of KB407 on pulmonary function, as measured by change from baseline in absolute and percent predicted FEV1 | 2 months
  Assessment of forced expiratory volume, in one second (FEV1,) will be assessed by spirometry as compared to baseline

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Gainesville, Florida
  - The Cystic Fibrosis Institute, Northfield, Illinois
  - New York Medical College/ Boston Children's Health Physicians, Hawthorne, New York
  - Northwell Health Physicians, New York, New York
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina